CLINICAL TRIAL: NCT04307498
Title: Predicting Treatment Outcomes With Intensive Outpatient Treatment for Posttraumatic Stress Disorder
Brief Title: Predicting Treatment Outcomes With Intensive Outpatient Treatment for PTSD
Acronym: PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Robert W. Woodruff Foundation (Other)
Responsible Party: Principal Investigator, Alan Peterson, Principle Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190788H
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2021-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Military; Veteran; Prolonged Exposure; Intensive Outpatient
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a prospective, one-group, exploratory clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intensive Outpatient Program - Prolonged Exposure (Other): Participants will complete fifteen weekday 90-minute Prolonged Exposure therapy sessions over three consecutive weeks plus seven augmentations designed to maximize treatment outcomes. If necessary, the treatment window may be extended for another week.
  Interventions: Behavioral: Intensive Outpatient Program - Prolonged Exposure

INTERVENTIONS:
Behavioral: Intensive Outpatient Program - Prolonged Exposure — Prolonged Exposure for Posttraumatic Stress Disorder (PE for PTSD; Foa, Hembree, & Rothbaum, 2007) is an empirically supported behavioral therapy that utilizes exposure-based interventions to target the psychological mechanisms (i.e., avoidance; maladaptive cognitive changes) thought to maintain trauma-related symptoms. IOP-PE includes 15 days of PE treatment delivered over three consecutive weeks. The standard outpatient PE protocol has modified with seven treatment augmentations to meet the unique needs of post-9/11 veterans.
  Other Names: IOP-PE

SUMMARY:
The open-label clinical study explores potential modifiable predictors of treatment outcomes in a sample of 55 military service members and veterans with clinically significant PTSD symptoms who receive Intensive Outpatient Prolonged Exposure (IOP-PE).

DETAILED DESCRIPTION:
Intensive Outpatient Prolonged Exposure (IOP-PE) is a three-week, intensive, individualized program that combines massed Prolonged Exposure with military-relevant treatment augmentations to treat posttraumatic stress disorder (PTSD; Peterson et al., 2018). Recent findings indicate that IOP-PE significantly decreased combat-related PTSD in post-9/11 service members and veterans (Peterson et al., 2019). However, IOP-PE is costly and requires a considerable commitment from the patient. Being able to prospectively identify which patients benefit most from IOP-PE will help treatment providers and patients make well-informed decisions about clinical care. The primary aim of this prospective, exploratory clinical study is to investigate potential predictors of treatment outcome following 15 sessions of IOP-PE delivered over 3-weeks in a sample of 55 military service members and veterans (i.e., individuals who have retired or separated from the US Armed forces, active duty personnel, reservists, and National Guardsmen/women) with significant PTSD symptoms. A follow-up assessment will be conducted one-month following the completion of treatment.

Predictor variables will include the following:

Aim 1: The PTSD Beliefs Inventory, the Dispositional Resilience and Disability Inventory, and the Credibility/ Expectancy Questionnaire.

Aim 2: The Disability-Recovery Implicit Association Test.

Aim 3: The Treatment Motivation Questionnaire and Service Connection Status

Aim 4: The Insomnia Severity Index, the Dimension of Anger Reactions-5, Patient Health Questionnaire-9, the Quick Drinking Screen, and the Pain Intensity, Enjoyment, and General Activity (PEG) Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military service members or veterans (18 years or older) who were impacted by Hurricane Harvey.
2. Significant PTSD symptoms as measured by a Posttraumatic Stress Disorder Checklist (PCL-5) score of 34 or higher.
3. Able to speak and read English (due to standardization of outcome measures)
4. Able to participate in a three-week intensive outpatient program

Exclusion Criteria:

1. Current manic episode or psychotic symptoms requiring immediate stabilization or hospitalization (as determined by the bipolar and psychosis modules of the Mini International Neuropsychiatric Interview (MINI) and clinical judgment)
2. Current and severe alcohol use warranting immediate intervention based on clinical judgment.
3. Evidence of a moderate or severe traumatic brain injury (as determined by the inability to comprehend the baseline screening questionnaires)
4. Current suicidal ideation severe enough to warrant immediate attention (as determined by the Depressive Symptoms Index - Suicidality Subscale and the Self-Injurious Thoughts and Behaviors Interview short form) and corroborated by a clinical risk assessment by a credentialed provider.
5. Other psychiatric disorders severe enough to warrant designation as the primary disorder as determined by clinician judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms | Baseline and 1 month follow-up
  Change in scale measurements by the Clinician Administered PTSD Scale (CAPS-5). The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Peterson, PhD, ABPP, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson AL, Foa EB, Blount TH, McLean CP, Shah DV, Young-McCaughan S, Litz BT, Schobitz RP, Castillo DT, Rentz TO, Yarvis JS, Dondanville KA, Fina BA, Hall-Clark BN, Brown LA, DeBeer BR, Jacoby VM, Hancock AK, Williamson DE, Evans WR, Synett S, Straud C, Hansen HR, Meyer EC, Javors MA, Sharrieff AM, Lara-Ruiz J, Koch LM, Roache JD, Mintz J, Keane TM; Consortium to Alleviate PTSD. Intensive prolonged exposure therapy for combat-related posttraumatic stress disorder: Design and methodology of a randomized clinical trial. Contemp Clin Trials. 2018 Sep;72:126-136. doi: 10.1016/j.cct.2018.07.016. Epub 2018 Jul 25. PMID 30055335
- [Background] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- See also: STRONG STAR website — http://www.strongstar.org